CLINICAL TRIAL: NCT06617858
Title: Open-label Phase 2 Trial of AMB-05X for Patients With ctDNA(+) Colorectal Cancer After Curative-intent Treatment
Brief Title: Trial of AMB-05X for Patients With ctDNA(+) Colorectal Cancer After Curative-intent Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0476; NCI-2024-07925 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMB-05X (Experimental)
  Interventions: Drug: AMB-05X

INTERVENTIONS:
Drug: AMB-05X — Given by IV

SUMMARY:
To investigate the efficacy of AMB-05X in patients with CRC with MRD as determined by a ctDNA(+) blood test and no clinically detectable radiographic disease.

DETAILED DESCRIPTION:
Primary Objective:

To determine ctDNA clearance rate at 6 months after treatment with AMB-05X in patients with stages I-IV CRC who have ctDNA(+) status after completion of standard of care, curative-intent therapies.

Exploratory Objectives:

To estimate 2-year DFS in patients with stage I-IV CRC with detectable ctDNA after completion of standard of care, curative-intent therapies) upon treatment with 6 months of AMB-05X.

To estimate 2-year OS in patients with stage I-IV CRC with detectable ctDNA after completion of standard of care, curative-intent therapies) upon treatment with 6 months of AMB-05X.

To determine the safety and tolerability of AMB-05X patients with stage I-IV CRC with detectable ctDNA after completion of standard of care, curative-intent therapies.

To characterize the pharmacokinetic profile of AMB-05X in patients with stage I-IV CRC who have ctDNA(+) MRD.

To correlate patterns of ctDNA change with clinical outcomes following treatment with AMB05X in patients with CRC who have detectable ctDNA after completion of standard therapies.

To associate clinical outcomes with PK, PD, anti-drug antibodies, and biomarkers obtained from tissue and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or pathologic confirmation of adenocarcinoma of the colon or rectum.
2. Completion of any curative intent therapies resulting in no evidence of disease (e.g., R0 resection) for stage I - IV CRC and has completed all planned adjuvant/standard therapies per the discretion of the evaluating clinician.
3. No evidence of measurable radiographic disease according to RECIST 1.1 criteria (Eisenhauer et al. Eur. J Cancer 2009) and/or clinically detectable disease (i.e., via endoscopy if utilized as part of standard of care assessment) at least 28 days after completion of all planned standard of care treatment.
4. A positive ctDNA assay (Signatera) at least 28 days after completion of all planned standard of care treatment. Assays performed at external institutions are accepted.
5. Adequate organ and marrow function as defined below:

   1. absolute neutrophil count: ≥1,000/mcL
   2. platelets: ≥75,000/mcL
   3. hemoglobin: .9.0 g/dL
   4. total bilirubin: ≤ institutional upper limit of normal (ULN)
   5. AST(SGOT)/ALT(SGPT): ≤1.5 × institutional ULN
   6. Creatinine clearance ≥50 mL/min. Creatinine clearance (CrCl) to be estimated by the Cockcroft-Gault equation as follows: Clcr (mL/min) = [(140 - age) x (weight in kg) ÷ [72 x (serum creatinine in mg/dL)] [0.85 if female]
6. ECOG performance status (PS) of 0 or 1 (Appendix A).
7. Age ≥ 18 years at the time of informed consent for study participation.
8. Ability to understand and willingness to sign a written informed consent document.
9. The effects of AMB-05X on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 90 days after the last dose of study treatment. (Refer to Pregnancy Assessment Policy

   MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.
10. Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
11. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of AMB-05X administration.

Exclusion Criteria:

1. Prior or concurrent malignancy within 3 years of registration whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen or requires concurrent therapy (examples include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, ductal carcinoma in situ, cervical carcinoma in situ).
2. Clinically significant hepatobiliary disease that, at the discretion of the treating investigator, would lead to excessive treatment risk on study.
3. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
4. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
5. Concomitant health conditions including, but not limited to, autoimmune or cardiovascular disorders that are deemed significant in the investigator's judgment.
6. Persistent adverse event greater than or equal to grade 2 of the Common Toxicity Criteria for Adverse Events (CTCAE) v.5.0 related to prior anti-cancer therapy (with the exceptions of alopecia and neuropathy).
7. Coexisting separate disease, metabolic disorder, clinically significant laboratory result, or any other condition that investigators suspect may (a) prohibit use of the investigational product, or (b) put the patient at undue risk of harm.
8. History of a grade 3 or 4 allergic reaction attributed to humanized or human monoclonal antibody therapy
9. Pregnant women are excluded from this study because AMB-05X is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AMB-05X, breastfeeding should be discontinued if the mother is treated with AMB-05X. These potential risks may also apply to other agents used in this study
10. Concurrent treatment with other systemic anti-cancer agents (e.g., chemotherapy, hormonal therapy, immunotherapy) or other treatments not part of protocol-specified anti-cancer therapy including concurrent investigational agents of any type.
11. Use of pexidartinib, any other oral tyrosine kinase inhibitor (e.g., imatinib or nilotinib), or any biologic treatment targeting CSF1 or CSF1R within the past 4 weeks.
12. Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Van Morris, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org